CLINICAL TRIAL: NCT04685278
Title: Anticardiolipin Autoantibodies as Useful Biomarker for the Prediction of Mortality in Septic Patients
Brief Title: Anticardiolipin Autoantibodies and Mortality in Septic Patients
Acronym: aCLsepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Military Hospital of Tunis (Other)
Responsible Party: Principal Investigator, Hajjej Zied, Professor, Military Hospital of Tunis
Other Study IDs: Military Hospital of Tunis
Record Dates: First submitted 2020-12-14; First posted 2020-12-28 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Morality
Keywords: anti-phospholipid; sepsis; intensive care unit
MeSH Terms: conditions — Sepsis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Blood samples — Blood samples were collected in dry tubes on days 1, 3, 5, 8 and 10 of hospitalization

SUMMARY:
The detection of antiphospholipid antibodies (aPL) is of interest because of their importance in the pathogenesis of arterial or venous thrombosis and their responsibility for a wide spectrum of clinical manifestations such as infection. The aim of the study was to assess the performance of antiphospholipid antibodies biomarker to predict in- hospital mortality in intensive care unit (ICU) septic patient's.

DETAILED DESCRIPTION:
the investigators conducted a prospective single-center observational study including consecutive critically ill septic adults admitted to the intensive care unit. Clinical and laboratory data including chemiluminescence immunoassay for antiphospholipid antibodies [anticardiolipin (aCL), antiphosphatidylserine (aPS)] were obtained. Blood samples were collected on days 1, 3, 5, 8 and 10 of hospitalization. The primary study endpoint was ICU mortality defined as death before ICU discharge. Secondary end points included correlation between SOFA score and biological parameters.

ELIGIBILITY:
Inclusion Criteria:

* patients, admitted to the ICU for sepsis and older than 18 years

Exclusion Criteria:

* pregnancy
* clinical history of antiphospholipid syndrome
* auto-immune diseases
* immunosuppressive treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients, admitted to the ICU for sepsis
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-02-05 (Estimated); Study Completion 2021-02-15 (Estimated)

PRIMARY OUTCOMES:
ICU mortality | mortality at day 14 of hospitalization
  Mortality was defined as death before ICU discharge Multivariate logistic regression modeling will beperformed to found factors associated with higher mortality

SECONDARY OUTCOMES:
correlation between SOFA score and antiphospholipid antibodies. | on days 1, 3, 5, 8 and 10 of hospitalization
  assess correlations between serum levels of both aCL and aPS and SOFA score

CONTACTS AND LOCATIONS:
Overall Officials: Iheb Labbene, Pr, Study Director — Military Hospital of Tunis
Locations (1):
- Military Hospital of Tunisia, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No